CLINICAL TRIAL: NCT00108914
Title: A Two Week Randomized, Double Blind Placebo Controlled, Parallel Group Study of GW685698X Aqueous Nasal Spray 100mcg and 50mcg QD in Pediatric Subjects With Perennial Allergic Rhinitis
Brief Title: Perennial Allergic Rhinitis Study In Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR30008
Record Dates: First submitted 2005-04-20; First posted 2005-04-21 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Perennial allergic rhinitis; pediatric
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

INTERVENTIONS:
Drug: GW685698X

SUMMARY:
The purpose of this study is to determine if the investigational drug is effective and safe in children with perennial allergic rhinitis.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Safety and Efficacy of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 50mcg and 100mcg for 12 Weeks in Pediatric Subjects Ages 2 to <12 Years with Perennial Allergic Rhinitis (PAR)

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of perennial allergic rhinitis.

Exclusion criteria:

* Have significant concomitant medical conditions.
* Use of corticosteroids or other allergy medications during the study.
* Have abnormal ECG.
* Have laboratory abnormality.
* Have abnormal eye exam.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 558 (Actual)
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Improvement in daily, reflective total nasal symptom scores after first 4-week treatment period in subjects ages 6 to <12 years.

SECONDARY OUTCOMES:
Improvement in AM, pre-dose, instantaneous total nasal symptom scores after first 4-week treatment period, overall evaluation of response to therapy for the first 4-week treatment period for subjects ages 6 to <12 years.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (60):
- United States (38):
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Cudahy, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Liverpool, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Bellevue, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, El Paso, Texas
- Argentina (4):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Finland (4):
  - GSK Investigational Site, Joensuu
  - GSK Investigational Site, Nokia
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Italy (6):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monticelli Ascoli Piceno
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Salerno
- Mexico (2):
  - GSK Investigational Site, México
  - GSK Investigational Site, Monterrey, N.L
- Slovakia (4):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Levoča
  - GSK Investigational Site, Nitra

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Máspero J, Rosenblut A, Finn A, J Lim J, Wu W, Philpot E. Safety of fluticasone furoate* nasal spray in children with perennial allergic rhinitis (*USAN approved name). Allergy 2007;62(Suppl. 83): 381 (abstract).
- [Result] Máspero JF, Rosenblut A, Finn A, Lim J, Wu W, Faris M, Philpot E. Once-daily fluticasone furoate nasal spray (FF) is safe and effective in the long-term treatment of perennial allergic rhinitis (PAR) in children ages 2 to 11 years. J Allergy Clin Immunol.
- [Result] Maspero JF, Rosenblut A, Finn A Jr, Lim J, Wu W, Philpot E. Safety and efficacy of fluticasone furoate in pediatric patients with perennial allergic rhinitis. Otolaryngol Head Neck Surg. 2008 Jan;138(1):30-7. doi: 10.1016/j.otohns.2007.10.023. PMID 18164990
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR30008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register